CLINICAL TRIAL: NCT01242371
Title: A Double-Blind Placebo-Controlled Trial of a Probiotic Supplement to Reduce the Symptoms of Schizophrenia
Brief Title: Double-Blind Trial of a Probiotic Supplement to Reduce the Symptoms of Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheppard Pratt Health System (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Faith Dickerson, Head, Stanley Research Program, Sheppard Pratt Health System
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SMRI/SPHS 2010-01
Record Dates: First submitted 2010-11-16; First posted 2010-11-17 (Estimated); Results first posted 2013-11-14 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-01

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Schizoaffective; Probiotic supplements; Gliadin; Casein
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotic Supplement (Active Comparator): Probiotic supplement 1 tablet by mouth daily for 14 weeks after 2 week placebo run-in
  Interventions: Dietary Supplement: Probiotic Supplement
- Identical-appearing Placebo (Placebo Comparator): Identical appearing placebo 1 tablet by mouth daily for 14 weeks after 2 week placebo run-in
  Interventions: Dietary Supplement: Identical-appearing Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic Supplement — Probiotic Supplement 1 tablet by mouth daily
  Arms: Probiotic Supplement
Dietary Supplement: Identical-appearing Placebo — Probiotic identical placebo 1 tablet by mouth daily
  Arms: Identical-appearing Placebo

SUMMARY:
The investigators intend to explore the hypothesis that symptoms of schizophrenia may be reduced by the administration of a probiotic supplement when used in addition to standard antipsychotic medications.

DETAILED DESCRIPTION:
The primary aim of the current study is:

1. To evaluate the safety and efficacy of a supplemental probiotic therapy, containing the microorganisms Lactobacillus rhamnosus GG and Bifidobacterium lanimalis subsp. lactis (BB12), for individuals with schizophrenia who have residual psychotic symptoms of at least moderate severity.

   Secondary aims of the study are:
2. To assess the effect of probiotic treatment on patients' gastrointestinal functioning
3. To study the effect of probiotic treatment in lowering the levels of antibodies to casein and gliadin.
4. To investigate the association between the efficacy of probiotic therapy and initial levels of antibodies to gliadin and casein.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65.
* Capacity for written informed consent.
* Primary Axis I diagnosis (DSM-IV) of schizophrenia, any type, OR schizoaffective disorder (APA, 1994).
* Currently an outpatient at the time of enrollment.
* Residual psychotic symptoms which are at least moderately severe as evidenced by one or more PANSS positive symptom scores, and/or PANSS negative symptom scores of 4 or more; OR a total PANSS score of 50 or more, containing at least three positive or negative items with scores of 3 or more at screening.
* Conformance to PORT Treatment Recommendation re Maintenance Antipsychotic Medication Dose (Buchanan et al., 2010).
* Receiving antipsychotic medication for at least 8 weeks prior to starting the study with no medication changes within the previous 21 days.
* Proficient in the English language.

Exclusion Criteria:

* Diagnosis of mental retardation.
* Any clinically significant or unstable medical disorder as determined by the investigators, including congestive heart failure, abnormal liver function or disease, renal failure, acute pancreatitis, any diagnosis of cancer undergoing active treatment, HIV infection or other immunodeficiency condition.
* History of IV drug use.
* Primary diagnosis of substance abuse or dependence according to DSM-IV criteria within the last three months.
* Participated in any investigational drug trial in the past 30 days.
* Pregnant or planning to become pregnant during the study period.
* Receipt of antibiotic medication within the previous 14 days (as anaerobic organisms residing in the gastrointestinal tract may be minimally affected by antibiotics).
* Documented celiac disease (as such persons should be on a gluten-free diet as this is the standard care).
* Of note, the investigators are not limiting the study to individuals with elevated levels of gliadin or casein antibodies as the investigators intend to look at these levels as a predictor of response.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2010-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Faith B Dickerson, PhD, MPH, Principal Investigator — Sheppard Pratt Health System
Locations (1):
- Sheppart Pratt Health System, Towson, Maryland, United States

REFERENCES:
- [Derived] Dickerson FB, Stallings C, Origoni A, Katsafanas E, Savage CL, Schweinfurth LA, Goga J, Khushalani S, Yolken RH. Effect of probiotic supplementation on schizophrenia symptoms and association with gastrointestinal functioning: a randomized, placebo-controlled trial. Prim Care Companion CNS Disord. 2014;16(1):PCC.13m01579. doi: 10.4088/PCC.13m01579. Epub 2014 Feb 13. PMID 24940526

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We enrolled n=65 participants drawn from rehabilitation and treatment programs in Central Maryland. Dates of recruitment 11/2010-01/2012.
Pre-assignment Details: We used a 2 week placebo run in for all participants prior to randomization. This placebo run in was followed by the 14 week double-blind treatment phase.
Groups:
- Probiotic Supplement: Probiotic supplement 1 tablet by mouth daily for 14 weeks
- Identical-appearing Placebo: Identical appearing placebo 1 tablet by mouth daily for 14 weeks
Period: Overall Study
Arm/Group | Probiotic Supplement | Identical-appearing Placebo
Started | 33 | 32
Completed | 31 | 27
Not Completed | 2 | 5
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Protocol Violation | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Probiotic Supplement | Identical-appearing Placebo | Total
Number analyzed (Participants) | 33 | 32 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 32 | 64
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (11.0) | 48.1 (9.4) | 46.2 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 23
  Male | 23 | 19 | 42
Region of Enrollment [Number; unit: participants]
  United States | 33 | 32 | 65

OUTCOME MEASURES:

1. Primary Outcome: Change in Positive and Negative Syndrome Scale (PANSS) Score From the Start to the End of the Double-blind Treatment Phase (Week 0 to Week 14)
Description: The Positive and Negative Syndrome Scale (PANSS) measures psychiatric symptomatology, especially related to psychosis. The complete PANSS contains ratings for 30 symptoms, including 7 positive symptoms, 7 negative symptoms, and 16 general psychiatric symptoms. The severity of each symptom is rated on a scale ranging from 1 (minimal) to 7 (extreme); higher scores indicate increased symptomatology. Total PANSS scores include scores from all categories and range from 30 to 210 units on a scale.
Time Frame: 14 weeks (week 0 to week 14)
Population: Week 0 data is based on the number of participants in the probiotic supplement group (n=33) and the placebo group (n=32) who began the treatment phase. Week 14 data is based on the number of participants in the probiotics supplement group (n=31) and the placebo group (n=27) who completed the treatment phase.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Probiotic Supplement | Identical-appearing Placebo
Number analyzed (Participants) | 33 | 32
units on a scale
  Wk 0 (Begin Treatment) PANSS Total Score, n=33,32 | 67.55 (11.64) | 69.56 (11.73)
  Wk 14 (End Treatment) PANSS Total Score, n=31,27: number analyzed (Participants) | 31 | 27
  Wk 14 (End Treatment) PANSS Total Score, n=31,27 | 67.42 (11.66) | 67.69 (11.86)

2. Secondary Outcome: Gastrointestinal Functioning From the Beginning to the End of the Double-blind Treatment Phase Weeks 0-14
Description: Self report rating of difficulty moving bowels on a 4 point scale from "no difficulty" to "severe difficulty"
Time Frame: 14 weeks (weeks 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13 & 14)
Reporting Status: Not Posted

3. Secondary Outcome: Measurement of Gliadin and Casein Antibody Levels
Time Frame: 16 weeks (baseline prior to placebo run in to week 14)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a 16 week period, including the 2 week placebo run in and the 14 week double-blind treatment phase.
Arm/Group | Probiotic Supplement | Identical-appearing Placebo
Serious Adverse Events (participants affected / at risk) | 2/33 | 1/32
Other Adverse Events (participants affected / at risk) | 19/33 | 21/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Probiotic Supplement (N=33) | Identical-appearing Placebo (N=32)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Schizophrenia exacerbation (Psychiatric disorders) | 2 (3) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Probiotic Supplement (N=33) | Identical-appearing Placebo (N=32)
Dermatological condition (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (6)
Diarrhea (Gastrointestinal disorders) | 9 (9) | 6 (8) — Diarrhea was assessed separately and is counted as a separate adverse event from other gastrointestinal problems, which were solicited non-specifically.
Gastrointestonal symptoms (excluding diarrhea) (Gastrointestinal disorders) | 5 (5) | 7 (9) — Non-specific new onset gastrointestinal symptoms including constipation, heartburn, nausea, stomach cramps, and/or flatulence. Diarrhea was assessed separately and is counted as a separate adverse event.
Genitourinary condition (Renal and urinary disorders) | 2 (2) | 2 (3)
Headache (Nervous system disorders) | 2 (3) | 1 (1)
Musculoskelatol condition (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Psychiatric condition (Psychiatric disorders) | 4 (4) | 2 (2) — Psychiatric disease under study
Upper respiratory illness (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 10 (10)

LIMITATIONS AND CAVEATS:
Did not perform more detailed measures of gastrointestinal functioning or obtain a more complete history of participants' gastrointestinal symptoms and associated treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No